CLINICAL TRIAL: NCT07324460
Title: One-Hour Positive Pressure Ventilation After a Pressure Support Spontaneous Breathing Trial: A Randomized Clinical Trial
Brief Title: One-Hour Positive Pressure Ventilation After a Pressure Support Spontaneous Breathing Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GS-Wean: PSV SBT
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Airway Extubation; Weaning Mechanical Ventilation; Extubation Failure
Keywords: Airway extubation; Weaning Mechanical Ventilation; Extubation failure
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-hour positive pressure ventilation (Experimental)
  Interventions: Other: One-hour positive pressure ventilation
- Immediate extubation (Active Comparator)
  Interventions: Other: Immediate extubation

INTERVENTIONS:
Other: One-hour positive pressure ventilation — As soon as the success of the spontaneous breathing trial is confirmed, the patient will be submitted to one-hour positive pressure ventilation using the previous ventilatory parameters and, afterwards, extubated.
  Arms: One-hour positive pressure ventilation
Other: Immediate extubation — The patient will be extubated immediately (up to 10 minutes) after the success of the spontaneous breathing trial.
  Arms: Immediate extubation

SUMMARY:
This is a randomized, open, multicenter, pragmatic, adaptive clinical trial with intention-to-treat analysis. The study will compare two weaning strategies from mechanical ventilation in critically ill patients admitted to intensive care units, with more than 72 hours of mechanical ventilation and with a successful spontaneous breathing trial on pressure support. Immediately after a successful spontaneous breathing trial, eligible patients will be randomized into 2 groups that will be treated according to one of the following interventions:1) One-hour positive pressure ventilation: as soon as the success of the spontaneous breathing trial is confirmed, the patient is submitted to mechanical ventilation for 1 hour using the previous ventilatory parameters and, afterwards, extubated.2) Immediate extubation: the patient is extubated immediately after the success of the spontaneous breathing trial.

DETAILED DESCRIPTION:
Adaptive design for sample size. The study will include up to a maximum of 4.000 patients. First interim analysis will be performed after complete data is available for the first 500 eligible patients. The Bayesian logistic regression model will be adjusted to provide posterior probabilities that will be compared with threshold values to evaluate stopping decisions. Extensive simulations were conducted to develop and understand adaptive design performance, interim analysis timing, and decision criteria. The trial may be stopped early for efficacy or futility. Secondary outcomes will be analyzed with a gatekeeping procedure to preserve overall type I error at 0.05. Thus, the assessment of statistical significance of secondary outcomes will be performed only if the preceding outcome in the hierarchy met the threshold for statistical significance. No adjustment for multiple comparisons will be applied for analyses of tertiary outcomes and subgroups. Thus, these results should be interpreted as exploratory.Secondary outcomes tested in hierarchical order will be: (1) Mechanical ventilation free days within 28 days; (2) Hospital free days within 28 days; (3) Mortality within 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years.
* Admitted to the intensive care unit (surgical or medical).
* With endotracheal intubation.
* Mechanical ventilation for more than 72 hours.
* Who underwent successful spontaneous breathing trial (according to the study protocol) and is considered able to be extubated.

Exclusion Criteria:

* Patients unable to obey commands.
* With non-planned extubation.
* Neuromuscular disease and cervical spinal cord injury.
* Tracheostomy.
* Contraindication for cardiopulmonary resuscitation or reintubation.
* Terminal extubation.
* Lack of informed consent.
* Previously included in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Extubation Failure Within 7 Days | 7 days (from randomization through Day 7 after randomization)
  Extubation failure is defined as a composite endpoint of reintubation or death within 7 days after randomization

SECONDARY OUTCOMES:
Ventilator-Free Days Through Day 28 | 28 days (from randomization through Day 28 after randomization)
  Ventilator-free days are defined as the number of days alive and free from invasive mechanical ventilation from randomization through Day 28 after randomization. If a patient dies before day 28, the ventilator-free days will be counted as zero. If a patient is reintubated and returns to mechanical ventilation and later is extubated again and remains in unassisted breathing until day 28, the ventilator-free days will be counted from the end of the last period of assisted breathing until day 28. An invasive mechanical ventilation period of less than 24 hours for surgical purposes will count as 1 ventilator-free day. Patients discharged from the hospital in unassisted breathing before 28 days will be considered alive and free from mechanical ventilation for the remaining days up to 28 days. Patients transferred to another hospital or healthcare unit will be followed up until day 28 to assess this outcome.
Hospital-Free Days Through Day 28 | 28 days (from randomization through Day 28 after randomization)
  Hospital-free days are defined as the number of days alive and out of the hospital from randomization through Day 28 after randomization. If a patient dies before day 28, the hospital-free days will be counted as zero. Patients discharged from the hospital in unassisted breathing before 28 days will be considered alive and free from hospital for the remaining days up to 28 days. Patients transferred to another hospital or healthcare unit will be followed through day 28 to ascertain this outcome.
Number of Participants Who Died Within 28 Days | 28 days (from randomization through Day 28 after randomization)
  All-cause mortality from randomization through day 28

OTHER OUTCOMES:
Ventilatory Support-Free Days Through Day 28 | 28 days (from randomization through Day 28 after randomization)
  Ventilatory support-free days are defined as the number of days alive and free from any ventilatory support (invasive or noninvasive) from randomization through day 28. Any use of invasive mechanical ventilation for any duration during a calendar day will count as 1 day with ventilatory support (i.e., not free). Use of noninvasive ventilatory support (noninvasive ventilation or high-flow nasal cannula) for ≥6 hours in any calendar day will count as 1 day with ventilatory support. Participants who die before day 28 will be assigned 0 ventilatory support-free days. If reintubation occurs and the participant later achieves unassisted spontaneous breathing again, ventilatory support-free days will be counted from the end of the last assisted-breathing period through day 28, provided the participant remains alive and free from ventilatory support.
Number of Participants With Extubation Failure Within 2 Days | 2 days (from randomization through Day 2 after randomization)
  Extubation failure is defined as a composite endpoint of reintubation or death within 2 days after randomization
Number of Participants With Death or Reintubation Within 28 Days | 28 days (from randomization through Day 28 after randomization)
  Composite endpoint of reintubation or death within 28 days after randomization
Intensive Care Unit-Free Days Through Day 28 | 28 days (from randomization through Day 28 after randomization)
  ICU-free days are defined as the number of days alive and out of the intensive care unit from randomization through day 28. If a patient dies before day 28, the ICU-free days will be counted as zero. Patients discharged from the hospital in unassisted breathing before 28 days will be considered as alive and free from ICU for the remaining days up to 28 days. Patients transferred to another hospital or healthcare unit will be followed up until day 28 to assess this outcome.
Number of Participants Who Died in the Intensive Care Unit | From randomization to ICU discharge, up to 90 days
  All-cause mortality occurring from randomization until ICU discharge (death before ICU discharge)
Number of Participants Who Died in the Hospital | From randomization to hospital discharge, up to 90 days
  All-cause mortality occurring from randomization until hospital discharge (death before hospital discharge)